CLINICAL TRIAL: NCT00360776
Title: A Phase 2 Study of Tipifarnib in Large Granular Lymphocyte (LGL) Leukemia
Brief Title: Tipifarnib in Treating Patients With Anemia or Neutropenia and Large Granular Lymphocyte Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00086; 5402; CDR0000489291; U01CA062502 (NIH); NCT00331591 (obsolete NCT alias)
Record Dates: First submitted 2006-08-03; First posted 2006-08-07 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Stage III Chronic Lymphocytic Leukemia; Stage IV Chronic Lymphocytic Leukemia; T-cell Large Granular Lymphocyte Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Large Granular Lymphocytic | interventions — tipifarnib

ARMS (1):
- Arm I (Experimental): Patients will receive tipifarnib by mouth twice a day for 3 weeks. Treatment may repeat every 4 weeks for up to eight courses.
  Patients will undergo blood collection periodically for laboratory studies. After finishing treatment, patients will be evaluated every 6 months for 5 years.
  Interventions: Drug: tipifarnib; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: tipifarnib — Given orally
  Other Names: R115777; Zarnestra
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well tipifarnib works in treating patients with anemia or neutropenia and large granular lymphocyte leukemia. Tipifarnib may stop the growth of leukemia by blocking blood flow to the cancer cells and by blocking some of the enzymes needed for cancer cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Estimate the complete response rate, partial response rate, and overall response rate in patients with natural killer (NK)- or T-cell-large granular lymphocyte (LGL) leukemia who present with neutropenia or anemia treated with tipifarnib.

SECONDARY OBJECTIVES:

I. Determine the toxicity of tipifarnib in these patients. II. Determine the mechanism of treatment responses in these patients through correlative laboratory studies.

OUTLINE: Patients are stratified by disease type (natural killer-large granular lymphocyte [LGL] leukemia vs T-cell-LGL leukemia).

Patients receive oral tipifarnib twice daily on days 1-21. Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients are evaluated after completion of course 4. Patients achieving complete response receive 1 additional course of treatment. Patients achieving partial response receive 4 additional courses of treatment in the absence of disease progression or unacceptable toxicity.

Patients undergo blood collection periodically during study for response mechanism studies and other biomarker correlative studies, including mutations of K-ras and N-ras genes.

After completion of study treatment, patients are followed every 6 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of T-cell-large granular lymphocyte (LGL) leukemia or natural killer (NK)-LGL leukemia associated with ≥ 1 of the following clinical manifestations:

  * Severe neutropenia (i.e., < 500/mm³)
  * Neutropenia associated with recurrent infections, meeting 1 of the following criteria: one severe infection requiring hospitalization or at least 2 infections requiring antibiotic therapy
  * Symptomatic anemia with significant fatigue with a score of greater than 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Status Scale; dyspnea on exertion, but able to walk one flight of stairs without stopping (less than grade 1 respiratory symptoms); cardiac symptoms including worsening of angina or new onset of chest pain
  * Transfusion-dependent anemia
* Willing to discontinue use of MTX, Cy, or cyclosporine for 1 month prior to study entry
* T-cell-LGL leukemia must meet all of the following criteria: CD3+ and CD57+ cells > 300/mm³ or CD8+ cells > 650/mm³ by phenotypic studies of peripheral blood, evidence for clonal T-cell receptor gene rearrangement based on positive flow cytometric analysis, T-cell receptor (TCR)-γ chain polymerase chain reaction (PCR), TCR-Vβ PCR, or by Southern blot analysis
* NK-LGL leukemia must have CD56+ or CD16+ NK cells > 750/mm³ by phenotypic studies of peripheral blood
* Life expectancy > 2 years
* ECOG performance status (PS) 0-2 OR Karnofsky PS 60-100%
* Fertile patients must use effective contraception prior to and during study
* Negative pregnancy test
* Normal kidney and liver function, as determined by the following laboratory results: total bilirubin less than or equal to 2.0 mg/dl; AST (SGOT) and ALT (SGPT) less than or equal to 2.5 times the upper limit of normal; and creatinine less than or equal to 2.0 mg/dl

Exclusion Criteria:

* Not pregnant or nursing
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to tipifarnib
* No allergies to imidazoles (e.g., clotrimazole, ketoconazole, miconazole, econazole, fenticonazole, isoconazole, sulconazole, tioconazole, or terconazole)
* No uncontrolled concurrent illness including, but not limited to, any of the following: ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, psychiatric illness or social situations that would limit study compliance
* No other serious medical illness that would limit survival to < 2 years
* No other malignancy within the past 5 years except inactive nonmelanoma skin cancer or carcinoma in situ of the cervix
* Psychiatric illness that may interfere with study participation
* No other anticancer agents or therapies
* No concurrent antiretroviral therapy for HIV-positive patients
* No other concurrent investigational agents
* No prior tipifarnib or other inhibitors of MAPK signaling intermediates

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-06-02 (Actual); Primary Completion 2007-05-14 (Actual)

PRIMARY OUTCOMES:
Response rates to tipifarib defined as the proportion of patients achieving a complete response (CCR) or partial response (PR) | Up to 5 years

SECONDARY OUTCOMES:
Changes in Ras/ERK and NK receptor expression | Baseline to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Loughran, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States